CLINICAL TRIAL: NCT02040935
Title: HOMERUS: A Local, Open Label, Multicentre, Phase IIIB Study, Investigating Subcutaneous Trastuzumab Administered at Home With Single Injection Device in Patients With HER2-Positive Early Breast Cancer
Brief Title: A Study of SC Administration of Trastuzumab (Herceptin) by SID at Home in HER2-Positive EBC Participants
Acronym: HOMERUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28878; 2013-000829-31 (EudraCT Number)
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (1):
- Trastuzumab (Experimental): Participants will receive 600 milligrams (mg) trastuzumab SC by SID every 3 weeks (Q3W) for up to a total of 1 year, unless disease recurrence, unacceptable toxicity or participant withdrawal occurs. The first 3 administrations will be done at hospital, after that participants will be permitted to self-administer under the supervision of a healthcare professional (HCP).
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — 600 mg SC Q3W by SID
  Other Names: Herceptin

SUMMARY:
This single-arm, open-label, local multicenter study will evaluate the safety and tolerability of trastuzumab administered subcutaneously (SC) by a single-use injection device (SID) in participants with human epidermal growth factor receptor 2 (HER2)-positive early breast cancer (EBC), following surgery and chemotherapy (neo-adjuvant or adjuvant).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast
* HER2-positive disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hormonal therapy will be allowed as per institutional guidelines
* Prior use of anti-HER2 therapy will be allowed
* Left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 50 percent (%)
* No evidence of residual, locally recurrent or metastatic disease after completion of surgery and chemotherapy, or during concurrent chemotherapy (neo-adjuvant or adjuvant)
* Use of concurrent radiotherapy will be permitted
* Completion of surgery and chemotherapy (if applicable)

Exclusion Criteria:

* History of other malignancy, except for participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma and participants with other curatively treated malignancies who have been disease-free for the last 5 years
* Participants with severe dyspnea at rest or requiring supplementary oxygen therapy
* Participants with other concurrent serious diseases that might interfere with planned treatment, including severe pulmonary conditions/illness
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab, specifically: history of documented congestive heart failure, high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), poorly controlled hypertension
* Pregnant or lactating women
* Women of childbearing potential and male participants with female partners of childbearing potential who are unable or unwilling to use adequate contraceptive methods during study treatment
* Concurrent enrollment in another clinical trial using an investigational anti-cancer treatment, including hormonal therapy, biphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any excipients of Herceptin, including hyaluronidase, or the adhesive of the SC device, or a history of severe allergic or immunological reactions, e.g. difficult to control asthma
* Inadequate hepatic or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | From Baseline up to approximately 4 years

SECONDARY OUTCOMES:
Pharmacokinetics: Trough Concentrations (Ctrough) of Trastuzumab | Pre-dose (within 1 day before trastuzumab administration) at Cycles 2, 3, 9, and 10, 12 or 13 (cycle length=21 days)
Health Survey Short Form-36 (SF-36) Score | Cycles 3 and 9 (cycle length=21 days)
Mood and Anxiety Questionnaire (MASQ) Score | Cycles 3 and 9 (cycle length=21 days)
Percentage of Participants Choosing to Return to Hospital Administration | Cycle 6 (cycle length=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Netherlands (17):
  - Medisch Centrum Alkmaar, Alkmaar
  - Meander Medisch Centrum; Locatie Lichtenberg, Amersfoort
  - Amphia ziekenhuis, locatie langendijk, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis; Oncology, Delft
  - Ziekenhuis Gelderse Vallei; Inwendige Geneeskunde, Ede
  - Martini Ziekenhuis, Groningen
  - Kennemer Gasthuis, Haarlem
  - Ziekenhuisgroep Twente, Hengelo, Hengelo
  - Tergooiziekenhuizen, loc. Hilversum, Hilversum
  - Spaarne Ziekenhuis Haarlem; Oncologie, Hoofddorp
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Franciscus Ziekenhuis, Roosendaal
  - Zuyderland ziekenhuis locatie Geleen, Sittard-Geleen
  - Haga Ziekenhuis, The Hague
  - VieCuri - Medisch Centrum voor Noord-Limburg, Venlo
  - Isala Klinieken, Zwolle